CLINICAL TRIAL: NCT06144073
Title: The Effect of Mandala Art Therapy in Coping With Premenstrual Syndrome: A Randomized Controlled Study
Brief Title: The Effect of Mandala Art Therapy in Coping With Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra KARATAŞ OKYAY, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSUESRAKARATASOKYAY002
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2023-11

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; Cope; Stress; Depression; Mandala
MeSH Terms: conditions — Premenstrual Syndrome; Depression | interventions — Methods; Population Groups

STUDY DESIGN:
Intervention Model Description: Intervention group (Mandala art therapy group) Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Mandala art therapy) group (Experimental): Students with premenstrual syndrome who were included in the mandala art therapy group by randomization method will be made to practice mandala.
  Interventions: Behavioral: Intervention (Mandala art therapy) group
- Control (No Intervention): Control group is the group without any intervention.

INTERVENTIONS:
Behavioral: Intervention (Mandala art therapy) group — Personal Information Form, Premenstrual Syndrome Scale, Coping with Premenstrual Change Scale, Perceived Stress Scale, Beck Depression Inventory will be applied to the students in both groups before mandala art therapy. The students in the experimental group will be given mandala activity by the researcher two days a week for 12 weeks/total 24 times. Three months after the first interview, Premenstrual Syndrome Scale, Coping with Premenstrual Change Scale, Perceived Stress Scale, Beck Depression Inventory will be administered as a post-test. One month after the end of the study, Premenstrual Syndrome Scale, Coping with Premenstrual Change Scale, Perceived Stress Scale, Beck Depression Inventory will be applied again as follow-up evaluation.
  Arms: Intervention (Mandala art therapy) group

SUMMARY:
Mandala practice will be applied to women with premenstrual syndrome. The intervention group (Mandala practice group) and the control group each consisted of 60 women.

DETAILED DESCRIPTION:
Materials and Methods: The randomized controlled trial was conducted between October 2022 and April 2024 with 120 students (60 intervention group and 60 control group) studying at Kahramanmaraş Sütçü İmam University and Gaziantep Islamic Science and Technology University, Faculty of Health Sciences, Department of Midwifery. In the study, mandala art therapy is applied to the students in the intervention group. The students will be informed about the method to be followed in the research, the voluntary information form will be read to those who want to participate in the research, and their verbal and written permission will be obtained. Before the mandala art therapy, Personal Information Form, Premenstrual Syndrome Scale (PMSS), Coping with Premenstrual Change Scale, Perceived Stress Scale, Beck Depression Inventory will be applied to the students in both groups. The students in the intervention group will be given mandala activity by the researcher two days a week for 12 weeks/total 24 times. Three months after the first interview, Premenstrual Syndrome Scale (PMSÖ), Coping with Premenstrual Change Scale, Perceived Stress Scale, Beck Depression Inventory will be administered as a post-test. One month after the end of the study, Premenstrual Syndrome Scale (PMS), Coping with Premenstrual Change Scale, Perceived Stress Scale, Beck Depression Inventory will be administered again as follow-up assessment. The materials such as drawing paper, drawing and crayons required for mandala drawing in the study were provided by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Having a regular menstrual history between 21-35 days
* Score above 110 on the PMSÖ
* Not taking medical treatment for PMS,
* No history of psychiatric illness,
* No gynecological disease,
* No recent use of antidepressants, benzodiazepines/antipsychotics, combined oral contraceptives or hormones,
* Volunteering to participate in the study.
* Not having received mandala art therapy training before,
* Not having a physical problem that would prevent mandala production,
* Active use of hands,
* No communication problems,
* Speaking Turkish,
* Suitability/willingness to work in a group.

Exclusion Criteria:

* Having a diagnosis of psychiatric illness
* Having a diagnosis of chronic disease
* History of drug use
* Under 18 years of age
* Unable to communicate verbally,
* Giving birth in the last 3 months or breastfeeding,
* Pregnant,
* Have a history of psychiatric illness (diagnosis of moderate or severe depression, psychosis, bipolar illness, eating disorder, somatic symptom disorder, or acute suicidality),
* Gynecological disease (e.g. hysterectomy, oophorectomy, gynecological cancer, polycystic ovary syndrome, infertility, endometriosis)
* Recent use of antidepressants, benzodiazepines/antipsychotics, combined oral contraceptives or hormones,
* Having a physical problem that prevents you from creating a mandala,
* The student has a physical disability in the upper extremity,
* Previous mandala art therapy training

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Determining the level of premenstrual syndrome | At the first interview, the Premenstrual Syndrome Scale was applied to all students in both groups as a pre-test.
  It is a five-point Likert-type scale consisting of 44 questions measuring the severity of premenstrual symptoms. The scale has a total of nine sub-dimensions including Depressive Affect, Anxiety, Fatigue, Irritability, Depressive Thoughts, Pain, Appetite Changes, Sleep Changes, and Bloating. The application of the premenstrual syndrome scale is carried out by retrospectively evaluating the person by taking into account the status of "being within one week before menstruation". "PMSQ Total Score" is obtained from the sum of the scores obtained from all sub-dimensions. A minimum of 44 and a maximum of 220 points can be obtained from the scale. An increase in the score indicates an increase in the intensity of PMS symptoms.
Determining the level of premenstrual syndrome | Three months after the first interview, the Premenstrual Syndrome Scale is administered as a pre-test to all students in both groups.
  It is a five-point Likert-type scale consisting of 44 questions measuring the severity of premenstrual symptoms. The scale has a total of nine sub-dimensions including Depressive Affect, Anxiety, Fatigue, Irritability, Depressive Thoughts, Pain, Appetite Changes, Sleep Changes, and Bloating. The application of the premenstrual syndrome scale is carried out by retrospectively evaluating the person by taking into account the status of "being within one week before menstruation". "PMSQ Total Score" is obtained from the sum of the scores obtained from all sub-dimensions. A minimum of 44 and a maximum of 220 points can be obtained from the scale. An increase in the score indicates an increase in the intensity of PMS symptoms.
Determining the level of premenstrual syndrome | One month after the post-test, the Premenstrual Syndrome Scale is administered to all students in both groups as a follow-up assessment.
  It is a five-point Likert-type scale consisting of 44 questions measuring the severity of premenstrual symptoms. The scale has a total of nine sub-dimensions including Depressive Affect, Anxiety, Fatigue, Irritability, Depressive Thoughts, Pain, Appetite Changes, Sleep Changes, and Bloating. The application of the premenstrual syndrome scale is carried out by retrospectively evaluating the person by taking into account the status of "being within one week before menstruation". "PMSQ Total Score" is obtained from the sum of the scores obtained from all sub-dimensions. A minimum of 44 and a maximum of 220 points can be obtained from the scale. An increase in the score indicates an increase in the intensity of PMS symptoms.
Identifying Coping with Premenstrual Change | At the first interview, the Coping with Premenstrual Change Scale was applied to all students in both groups as a pre-test.
  "Coping with Premenstrual Change Scale (PMS-Coping)" It has 17 items and three sub-dimensions (Seeking Positive Affecting Behaviors, Seeking Support, Health Care Utilization Behavior). The items of the scale are answered on a 4-point Likert scale. The scale includes the options of "strongly disagree" (1 point), "not sure" (2 points), "agree" (3 points) and "strongly agree" (4 points). The minimum score is 17 and the maximum score is 68. In the instructions of the scale, it is asked to answer by thinking about the days before menstruation starts. The scale is used to describe the methods used to cope with premenstrual change in women.
Identifying Coping with Premenstrual Change | Three months after the first interview, the Coping with Premenstrual Change Scale is administered as a pre-test to all students in both groups.
  "Coping with Premenstrual Change Scale (PMS-Coping)" It has 17 items and three sub-dimensions (Seeking Positive Affecting Behaviors, Seeking Support, Health Care Utilization Behavior). The items of the scale are answered on a 4-point Likert scale. The scale includes the options of "strongly disagree" (1 point), "not sure" (2 points), "agree" (3 points) and "strongly agree" (4 points). The minimum score is 17 and the maximum score is 68. In the instructions of the scale, it is asked to answer by thinking about the days before menstruation starts. The scale is used to describe the methods used to cope with premenstrual change in women.
Identifying Coping with Premenstrual Change | One month after the post-test, the Coping with Premenstrual Change Scale is administered to all students in both groups as a follow-up assessment.
  "Coping with Premenstrual Change Scale (PMS-Coping)" It has 17 items and three sub-dimensions (Seeking Positive Affecting Behaviors, Seeking Support, Health Care Utilization Behavior). The items of the scale are answered on a 4-point Likert scale. The scale includes the options of "strongly disagree" (1 point), "not sure" (2 points), "agree" (3 points) and "strongly agree" (4 points). The minimum score is 17 and the maximum score is 68. In the instructions of the scale, it is asked to answer by thinking about the days before menstruation starts. The scale is used to describe the methods used to cope with premenstrual change in women.

SECONDARY OUTCOMES:
Determination of Perceived Stress Level | At the first interview, the Perceived Stress Level Scale was applied to all students in both groups as a pre-test.
  The Perceived Stress Level Scale (PSL) consists of 14 items. It was created to measure the extent to which people perceive certain situations in their lives as stressful. The scale is a 5-point Likert-type scale (0: Never, 1: Almost Never, 2: Sometimes, 3: Frequently, 4: Very often). The questions in the scale are aimed at evaluating the change in the participants' emotional state in the last one month. The stress level perceived by the respondent is determined by summing the scores obtained from the items. The scale has a total score between 0-56 points and the higher the score, the higher the perceived stress level.
Determination of Perceived Stress Level | Three months after the first interview, the Perceived Stress Level Scale is administered as a pre-test to all students in both groups.
  The Perceived Stress Level Scale (PSL) consists of 14 items. It was created to measure the extent to which people perceive certain situations in their lives as stressful. The scale is a 5-point Likert-type scale (0: Never, 1: Almost Never, 2: Sometimes, 3: Frequently, 4: Very often). The questions in the scale are aimed at evaluating the change in the participants' emotional state in the last one month. The stress level perceived by the respondent is determined by summing the scores obtained from the items. The scale has a total score between 0-56 points and the higher the score, the higher the perceived stress level.
Determination of Perceived Stress Level | One month after the post-test, the Perceived Stress Level Scale is administered to all students in both groups as a follow-up assessment.
  The Perceived Stress Level Scale (PSL) consists of 14 items. It was created to measure the extent to which people perceive certain situations in their lives as stressful. The scale is a 5-point Likert-type scale (0: Never, 1: Almost Never, 2: Sometimes, 3: Frequently, 4: Very often). The questions in the scale are aimed at evaluating the change in the participants' emotional state in the last one month. The stress level perceived by the respondent is determined by summing the scores obtained from the items. The scale has a total score between 0-56 points and the higher the score, the higher the perceived stress level.
Determination of Depression Level | At the first interview, the Beck Depression Inventory was applied to all students in both groups as a pre-test.
  The Depression Inventory consists of 21 items, 15 of which include psychological and 6 somatic symptoms. Although the inventory is a 4-point Likert-type inventory (scored between 0-3), it is used in various researches and clinical applications. The highest score that can be obtained from the inventory is 63 and the lowest score is 0. A high total score indicates a high level of depression. The cut-off point for clinical significance of depression is 17 points.
Determination of Depression Level | Three months after the first interview, the Beck Depression Inventory is administered as a pre-test to all students in both groups.
  The Depression Inventory consists of 21 items, 15 of which include psychological and 6 somatic symptoms. Although the inventory is a 4-point Likert-type inventory (scored between 0-3), it is used in various researches and clinical applications. The highest score that can be obtained from the inventory is 63 and the lowest score is 0. A high total score indicates a high level of depression. The cut-off point for clinical significance of depression is 17 points.
Determination of Depression Level | One month after the post-test, the Beck Depression Inventory is administered to all students in both groups as a follow-up assessment.
  The Depression Inventory consists of 21 items, 15 of which include psychological and 6 somatic symptoms. Although the inventory is a 4-point Likert-type inventory (scored between 0-3), it is used in various researches and clinical applications. The highest score that can be obtained from the inventory is 63 and the lowest score is 0. A high total score indicates a high level of depression. The cut-off point for clinical significance of depression is 17 points.

CONTACTS AND LOCATIONS:
Overall Officials: Esra KARATAŞ OKYAY, Principal Investigator — Kahramanmaras Sutcu Imam University; Zeynep BAL, PhD, Study Director — Gaziantep Islam Science and Technology University; Hatice POLAT, PhD, Study Director — Malatya Turgut Ozal University
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziantep Islamic University of Science and Technology, Gaziantep
  - Kahramanmaras Sutcu Imam University, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Background] Jang SH, Kim DI, Choi MS. Effects and treatment methods of acupuncture and herbal medicine for premenstrual syndrome/premenstrual dysphoric disorder: systematic review. BMC Complement Altern Med. 2014 Jan 10;14:11. doi: 10.1186/1472-6882-14-11. PMID 24410911
- See also: Description citation link — https://pubmed.ncbi.nlm.nih.gov/24410911/